CLINICAL TRIAL: NCT07199296
Title: A Prospective, Multicenter, Open-Label Clinical Study of Orelabrutinib in Combination With Rituximab With Optional Autologous Hematopoietic Stem Cell Transplantation in Treatment-Naive, Non-High-Risk Mantle Cell Lymphoma (MCL)
Brief Title: Orelabrutinib and Rituximab With Optional Autologous Hematopoietic Stem Cell Transplantation in MCL Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Qilu Hospital of Shandong University (Other); Huadong Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OR+/-ASCT
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib; Rituximab; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Orelabrutinib + Rituximab +/- ASCT and Orelabrutinib Maintenance (Experimental): 1. In induction phase, patients will receive rituximab 375 mg/m² IV on day 1,8,15,22 in Cycle 1, then day 1/cycle, and orelabrutinib 150 mg/day PO once daily, every 28 day per cycle for 6 cycles. Patients with an objective response (complete or partial) after induction therapy, who meet ASCT eligibility criteria and consent, proceed to transplantation.
  2. ASCT: BEAM pretreatment. Patients receive carmustine on day -7, etoposide on days -6-(-3), cytarabine on days -6-(-3) and melphalan on day -2.
  3. In maintenance phase, patients will recieve orelabrutinib 150 mg/day PO once daily until disease progression or intolerable toxicity.
  Interventions: Drug: Orelabrutinib; Drug: Rituximab (R); Drug: BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan); Drug: orelabrutinib maintenance

INTERVENTIONS:
Drug: Orelabrutinib — orelabrutinib 150mg/day PO once daily
  Other Names: Induction phase
Drug: Rituximab (R) — rituximab 375 mg/m² IV on day 1, 8, 15, 22 in Cycle 1, then day 1/cycle
  Other Names: Induction phase
Drug: BEAM (carmustine (BCNU), etoposide, cytarabine, melphalan) — the reference doses are as follows (each center may adjust them as appropriate based on actual conditions): carmustine 300mg/m² IV d-1; etoposide 200mg/m² IV d-6-(-3); cytarabine 200mg/m² IV d-6-(-3); melphalan 140mg/m² IV d-2.
Drug: orelabrutinib maintenance — orelabrutinib 150mg/day PO once daily

SUMMARY:
This multicenter, open-label, trial aims to evaluate the efficacy and safety of orelabrutinib in combination with rituximab with optional autologous hematopoietic stem cell transplantation in patients with non-high-risk mantle cell lymphoma (MCL). The primary objective is to assess the optimal complete response (CR) rate during the induction phase, with secondary objectives including progression-free survival (PFS), overall survival (OS), objective response rate (ORR), and safety. Exploratory analysis will investigate the correlation between tumor biomarkers and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MCL (mantle cell lymphoma) through flow cytometry or histopathology, and has not received prior treatment.
* Age > 14 years of age, both genders are eligible.
* Ann Arbor stage II-IV; for stage II subjects, those who require systemic therapy based on the investigator's judgment are eligible.
* At least one measurable lesion.
* Laboratory tests (blood routine, liver and kidney function) meet the following requirements: a) Blood routine: White blood cell count ≥3.0×10^9/L, absolute neutrophil count ≥1.5×10^9/L, hemoglobin ≥90g/L, platelet count ≥75×10^9/L. b) Liver function: Transaminases ≤2.5 times the upper limit of normal, bilirubin ≤1.5 times the upper limit of normal. c) Serum creatinine 44-133 mmol/L.
* The investigator judges that the subject's life expectancy is greater than 12 weeks from the time of screening.
* Willing and able to participate in all required assessments and procedures of the study protocol.

Exclusion Criteria:

* Patients who have previously received treatment with BTK inhibitors.
* Any one of the following high-risk factors is present: MIPI score of 6-11, Ki67 > 30%, TP53 abnormality, blastic or pleomorphic variation.
* Patients with severe complications or serious infections.
* Patients with uncontrolled cardiovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.
* Patients with active infections requiring systemic treatment, including bacterial, fungal, and viral infections.
* HIV-infected individuals.
* Patients with mental disorders or those who are known or suspected to be unable to fully comply with the study protocol.
* Patients whom the investigator judges to have other conditions that make them unsuitable for participation in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall Response Rate | End of induction treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=28 days]
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | Baseline up to data cut-off (up to approximately 3 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 3 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No